CLINICAL TRIAL: NCT07347405
Title: A Randomized Double-masked Dose-controlled Trial to Assess the Tolerability, Safety, Subjective Experience, and Efficacy of Repeated Administration of Three Different Doses of Psilocybin Whole Mushroom for the Treatment of Obsessive-compulsive Disorder.
Brief Title: Psilocybin Whole Mushroom for the Treatment of Obsessive-compulsive Disorder.
Acronym: Mushroom-OCD
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Francisco A Moreno (Other)
Collaborators: Arizona Biomedical Research Commission (ABRC) (Other)
Responsible Party: Sponsor-Investigator, Francisco A Moreno, MD, Professor of Psychiatry, University of Arizona
Organization: University of Arizona (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 00005573
Record Dates: First submitted 2025-12-22; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose 10 mg (Experimental): Whole dried psilocybin mushroom containing 10 mg of psilocybin will be mixed in a chocolate matrix and administered to the patient.
  Interventions: Drug: Psilocybin 10 mg
- Middle dose 20 mg (Experimental): Whole dried psilocybin mushroom containing 20 mg of psilocybin will be mixed in a chocolate matrix and administered to the patient.
  Interventions: Drug: Psilocybin 20 mg
- High dose 30 mg (Experimental): Whole dried psilocybin mushroom containing 30 mg of psilocybin will be mixed in a chocolate matrix and administered to the patient.
  Interventions: Drug: Psilocybin 30 mg

INTERVENTIONS:
Drug: Psilocybin 10 mg — Oral administration of whole dried psilocybin mushrooms contained in a chocolate matrix.
  Arms: Low dose 10 mg
Drug: Psilocybin 20 mg — Oral administration of whole dried psilocybin mushrooms contained in a chocolate matrix.
  Arms: Middle dose 20 mg
Drug: Psilocybin 30 mg — Oral administration of whole dried psilocybin mushrooms contained in a chocolate matrix.
  Arms: High dose 30 mg

SUMMARY:
The study tries to improve our treatments for people who have obsessive-compulsive disorder (OCD) by testing psilocybin, a mind altering drug that changes activity in brain areas involved in OCD. 30 patients with moderate or more severe OCD who are not taking mind altering medications or street drugs will participate in a 12 week study. Participants will be assigned (by luck of the draw) to take a low, medium, or high dose whole psilocybin mushroom contained in three chocolate pieces, prepared for this study by the Scottsdale Research Institute.

DETAILED DESCRIPTION:
Participants will come to the University of Arizona CATS Research Unit in Tucson for assessment, if they are found to be fit for study participation, they will be scheduled for a preparation session with a study therapist and then will participate in a dosing session when they will ingest three pieces of chocolate containing psilocybin mushroom. They will answer questions of how they are feeling, and will be monitored for safety by two study staff members, and their vital signs will be checked every hour on the day they receive the study drug. The will be sent home with a responsible adult selected by the patient after they are felt to be safe once the effects of the drug have resolved. Participants will receive four different doses separated by about three weeks. After they complete the treatment phase, they will be contacted monthly for follow up assessment of efficacy, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old, and older
* Have OCD (DSM-5) based on diagnostic interview using the Structured Clinical Interview for DSM-5 Research Version (SCID).
* At least moderate severity: Yale-Brown Obsessive Compulsive Scale (YBOCS) score ≥16.
* Failed at least one adequate trial of guideline concordant treatment.
* Considered safe for independent living
* Subjects must discontinue use of any of the following prescription or over the counter (OTC) products or nutritional supplements at least two weeks prior to initiating double-blind treatment:

  * Monoamine oxidase (MAOI), UGT1A10, and UGT1A9 inhibitors
  * Other active OCD treatments (cognitive behavioral therapy [CBT] or other psychotherapy; electrical or magnetic device treatments; pharmacological treatments such as antidepressant medications (e.g., SSRIs, SNRIs, MAOIs, TCAs, 5HT2 blockers, NERIs, etc.), lithium, antipsychotic drugs, 5-HT2 antagonists such as pimavanserin, and glutamatergic acting medications)

    * Note that fluoxetine must be discontinued at least 6 weeks prior to initiating double-blind treatment.
  * 5HT2 agonists (e.g., efavirenz, lorcaserin), which may alter the response to psilocybin
  * Serotonin-acting dietary supplements (e.g., 5-hydroxy-tryptophan, St. John's wort) due to potential for interaction with psilocybin and increased safety risks

Exclusion Criteria:

* Concurrent active substance use disorder, or a personal history of psychosis.
* History of psychosis among first degree relatives as determined by the Family Interview for Genetic Studies (FIGS)32
* Medical illness based on physical examination and routine blood testing that may complicate cardiovascular safety or drug metabolism or excretion. Examples include: 1) Cardiovascular conditions: lifetime history of stroke, lifetime myocardial infarction, uncontrolled hypertension (resting blood pressure >140/90 mmHg), tachycardia (resting heart rate >100 beats per minute), elongated QT interval corrected by Fridericia's formula (QTcF; interval >450 msec), participants with existing valvular heart disease, or clinically significant arrhythmia (<1 year prior to signing the ICF); 2) Metabolic conditions: subjects with diabetes should have a stable diabetes treatment regimen and no history of diabetic ketoacidosis, hyperglycemic coma, or no hypoglycemic episodes with glucose below 54 mg/dL in the 3 months prior to baseline, and fasting glucose >70 mg/dL at baseline; 3) Severe renal impairment: eGFR <45 mL/min/1.73 m²); and Liver failure: Child-Pugh Classes B and C.
* Unstable Chronic Obstructive Pulmonary Disease (COPD) or severe sleep apnea
* Clinically significant renal or hepatic impairment, per clinical judgment of a study physician
* EKG QTc ≥ 450 msec
* Psychiatric comorbidity that may represent an acute risk to their own or other's safety, including history of bipolar disorder (I or II) in the participant or first degree relative, as well as any family history of psychosis.
* Subjects cannot require any sedative, narcotic, or neuroleptic medications on a regular basis. Any of these medications they have taken should have been stopped long enough in the past to allow for their elimination and safe withdrawal prior to starting administration of the study drug. The specific time required will be dependent on the medication the patient was previously receiving.
* Participants who are pregnant, breastfeeding, planning a pregnancy, or planning to donate sperm within three months post-last study drug administration.
* Participants of childbearing potential or participants with partners of childbearing potential who engage in intercourse which could result in pregnancy are unwilling/unable to practice medically acceptable highly effective birth control (double barrier, oral and injectable pharmacological contraceptives, or surgical such as vasectomy or bilateral tubal occlusion) during the study and up to three months after the last study drug administration.
* Suicide attempt within the 12 months prior to enrollment
* Any condition for which MRI is contraindicated, at the discretion of a study investigator or the MRI technician, including: Pacemakers and defibrillators; artificial heart valves which are not MRI safe; any metal in head, spinal cord, eyes or chest; any electrical devices such as cochlear implants, nerve stimulators, deep brain stimulators, gastric pacemaker, or insulin or pain pumps; aneurysm clips; ferrous (i.e. non titanium alloy) implants in any part of the body.
* Use within the week prior to screening of drugs of abuse as listed in the current US DOJ DEA Drugs of Abuse Resource Guide, including:

  * Cannabinoids (marijuana, synthetic cannabinoids)
  * Simulants (amphetamine, cocaine, methamphetamine, methylphenidate, modafinil)
  * Opioids (natural and synthetic),
  * Sedatives (benzodiazepines, barbiturates, GHB, zolpidem, zaleplon, zopiclone)
  * Hallucinogens (DMT, ibogaine, LSD, MDMA, psilocybin, psilocin, PSP)
* Weight below 45kg
* Allergy or significant intolerance to chocolate or cocoa

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale | Baseline, Weekly for 12 weeks (Treatment phase), and Monthly for 12 month (Follow up phase).
  Clinician rating scale to determine severity of OCD symptoms. Scores vary from 0 to 40. Higher scores represent greater severity of OCD symptoms.
Adverse Event (AE) Tracking log | Weekly for 12 weeks (Treatment phase), and Monthly for 12 month (Follow up phase).
  The Adverse Event tracking log will collect information on adverse health events reported throughout the research study.
Visual Analogue Scale (VAS) | Baseline, Weekly for 12 weeks (Treatment phase), and Monthly for 12 month (Follow up phase). Scale 0 (no symptoms at all) to 100 (maximum symptom severity)
  Self-reported measure of intensity or frequency of pain or other various symptoms

SECONDARY OUTCOMES:
World Health Organization's quality of life assessment (WHOQOL-BREF) | Baseline, Weekly for 12 weeks (Treatment phase), and Monthly for 12 month (Follow up phase).
  A 26-item psychometric questionnaire to measure quality of life and functional ability. Raw scores are converted to transformed scores in four health related domains. Higher scores represent higher quality of life.
Short form health survey (SF-36) | Baseline, Weekly for 12 weeks (Treatment phase), and Monthly for 12 month (Follow up phase). Functionality scales are transformed to range from 0 to 100 with 0 being maximal disability and 100 being no disability.
  Subject self-reporting health survey to monitor and assess functional impairment
Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline, Weekly for 12 weeks (Treatment phase), and Monthly for 12 month (Follow up phase). Individuals with positive ideation or behavior scores can be categorized into low, moderate or high risk of suicide.
  A suicide risk assessment tool for prospective monitoring of suicidal ideation and behavior.

IPD SHARING:
Plan to Share IPD: No